CLINICAL TRIAL: NCT00742768
Title: Comparison of Absorption of Vitamin K2 Human Study Gelpell
Brief Title: Comparison of Absorption of Vitamin K2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: VitaK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 08-3-012
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2009-03

CONDITIONS: Healthy
Keywords: absorption; encapsulation; menaquinone; Bio-availability
MeSH Terms: interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): softgel capsules
  Interventions: Dietary Supplement: Vitamin K2 in softgel
- 2 (Active Comparator): Gelpell capsules
  Interventions: Dietary Supplement: Vitamin K2 in Gelpell

INTERVENTIONS:
Dietary Supplement: Vitamin K2 in softgel — 4 softgel capsules containing 45 µg MK-7 and 5 µg vitamin D3 per capsule and 4 softgel capsules containing 30 µg MK-4 per capsule
  Arms: 1
Dietary Supplement: Vitamin K2 in Gelpell — 4 Gelpell capsules containing 45 µg MK-7 and 5 µg vitamin D3 per capsule and 4 Gelpell capsules containing 30 µg MK-4 per capsule
  Arms: 2

SUMMARY:
From previous studies it appeared that menaquinone-7 (MK-7) is the most effective form of vitamin K. The Japanese soya product natto is one of the richest food sources of MK-7. However, the taste of natto is not appreciated by the western society. For this reason the active biological compound is produced as a capsule. Different techniques of encapsulation the vitamin can lead to different absorption profiles with intake. Therefore it is important to study influence of type of encapsulation technique on absorption of menaquinone-7.

This study is undertaken to compare absorption of menaquinones between two different encapsulation techniques. Absorption profiles of menaquinone-4 and menaquinone-7 of conventional softgel capsules and newly developed GellpelTM capsules are compared between each other.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 20 and 30 years old
* Subjects of normal body weight and height according to BMI < 30
* Subjects of Caucasian race
* Subject has given written consent to take part in the study

Exclusion Criteria:

* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects presenting chronic degenerative and/or inflammatory disease
* Subjects receiving corticoϊd treatment
* Subjects using oral anticoagulants
* Subject with (a history of) soy allergy
* Subjects using vitamin K containing multivitamins or vitamin K supplements
* Subjects with anaemia or subjects who recently donate blood.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The mean difference in plasma concentration of MK-4 and MK-7 between the two types of capsules (softgel or gelpell)concerns the primary outcome measure. | 4 weeks

SECONDARY OUTCOMES:
The mean difference in serum concentration of vitamin D3 between the two types of capsules (softgel or gelpell) concerns the secondary endpoint for this study. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — Maastricht University, VitaK BV
Locations (1):
- VitaK BV / Maastricht University, Maastricht, Netherlands